CLINICAL TRIAL: NCT01875588
Title: An Evaluation of HIV-associated Neurocognitive Disorders (HAND) in Virologically Controlled Patients
Brief Title: Thinking and Memory Problems in People With HIV
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130149; 13-N-0149
Record Dates: First submitted 2013-06-11; First posted 2013-06-12 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01-09

CONDITIONS: HIV Positive
Keywords: Healthy Controls; HIV Positive; Neuropyschological Testing; Thinking and Memory; Lumbar Drain/Puncture; Natural History
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DOD: Participants that are from IDCRP
- HIV negative controls: Participants that do not have HIV infection
- HIV positive: Participants that have HIV infection

SUMMARY:
Background:

- People with human immunodeficiency virus (HIV) can sometimes develop thinking and memory problems. These problems can vary widely, from few symptoms to severe problems with memory and concentration. It initially was thought that good HIV treatment could prevent almost all HIV-related memory problems. However, even people with low HIV viral loads can have these problems. It may be caused by HIV affecting the brain and spinal fluid. It is not yet clear why HIV causes these problems and why they may be worse in some people than others. Researchers want to study people with HIV and healthy volunteers to see how HIV may affect people with only small amounts of the virus in their blood.

Objectives:

- To study thinking and memory problems in individuals with HIV that is otherwise controlled with medications.

Eligibility:

* Individuals between 18 of age or older whose HIV has been controlled with medications for at least 1 year.
* Healthy volunteers between 18 of age or older.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. A neurological test will also be given. Participants will have a baseline imaging study of the brain.
* Within 12 weeks of the first visit, participants will have a second visit. Additional blood samples will be drawn. Another brain imaging study will be performed.
* Within 8 weeks of the second visit, participants will have a third visit to collect more blood samples. They will also provide spinal fluid samples, either as a single visit or a longer procedure.
* After this visit, participants will return every 12 months for up to 10 years. Blood samples will be collected as needed at these visits. Thinking and memory tests and imaging studies may also be given as needed. Spinal fluid may be collected at one visit a year.

DETAILED DESCRIPTION:
The natural history of neurocognitive impairment in human immunodeficiency virus (HIV)-infected individuals remains poorly understood. While the advent of highly active antiretroviral therapy (HAART) has led to a decreased incidence of the most severe form of HIV associated neurocognitive disorders (HAND), HIV-associated dementia, it does not appear to have impacted overall prevalence of HAND. Existing evidence suggests that the central nervous system (CNS) could be an important reservoir for HIV regardless of cumulative time on treatment. This 20 year multi-institute natural history protocol will identify approximately 500 HIV-infected individuals and 250 healthy volunteers for enrollment in multiple HAND studies at the National Institutes of Health (NIH). Participants will undergo a screening and evaluation assessment, which will include blood and urine collection, neuropsychological testing, Client Diagnostic Questionnaire (CDQ), and brain magnetic resonance imaging (MRI) with optional lumbar puncture and ophthalmology exam to repeat yearly for up to ten years.

The option to have a lumbar drain is only on the first visit and extended to HIV positive individuals only. Participants will have the option of doing a positron emission tomography/computed tomography (PET/CT) imaging if they have previously had a PET/CT scan under this study. Cerebrospinal fluid (CSF) markers of immune activation, chronic monocyte activation, cytomegalovirus/Epstein-Barr virus (CMV/EBV) infection/reactivation, and neuronal injury will be collected. In addition, HIV viral load and genotype, genetic susceptibility factors and CNS penetration-effectiveness score (CPE) and CSF levels of antiretroviral drugs may be assessed. A repository of cryopreserved biological samples will be developed and used for validation of candidate biomarkers in future studies. Collection and analysis of these data will not only enhance understanding of the CNS as a potential HIV reservoir in virally-controlled individuals but will further define the association among cortical thickness, biomarkers and neurocognitive function in an aging HIV-infected population.

ELIGIBILITY:
* INCLUSION CRITERIA:

All Participants (HIV-infected and HIV-negative Controls):

While different individual HIV neurocognitive studies have specific selection criteria, especially related to HIV viral load and antiretroviral therapy, inclusion criteria for this overarching protocol will be flexible in order to identify the broadest base of potential enrollees possible.

1. 18 years of age and older.
2. Ability to sign informed consent by the participant.
3. At least seventh grade educational level and ability to speak, read, and understand English. Education level will be assessed by participant self-report. Because many of the neuropsychological subtests were validated using United States norms, participants must be native English speakers or if foreign-born, demonstrate ability to understand the English language at the time of protocol consent and neuropsychological testing.
4. Consent to store blood and tissue.
5. Willing to participate in this study for up to 20 years.

HIV-infected Only:

1. HIV-1 infection, as documented by OraQuick rapid test using venipuncture whole blood, or fingerstick whole blood; or with HIV-1/HIV-2 Multispot rapid test and Western Blot as determined by NIH Clinical Pathology Laboratory or Leidos Biomedical Research. Monitoring Laboratory.
2. Outside primary medical doctor who provides care.
3. Plasma HIV-RNA <50 copies/mm3 or BLD for greater than one year. Participants who experience transitory episodes of an HIV viral load > 50 copies/mm3 preceded and followed by plasma viremia < 50 copies/mm3 may be included.
4. At least one year of continuous ART.

HIV-negative Controls Only:

1.HIV-antibody negative but can be taking pre-exposure prophylaxis (PrEP).

EXCLUSION CRITERIA:

1. Illness or other condition that, in the opinion of the PI, may interfere with study participation at the time of enrollment, including, but not limited to those listed below:

   1. CNS infections: this includes but is not limited to Varicella zoster virus (VZV) encephalitis, CNS lymphoma and toxoplasmosis. Participants who have recovered from effectively treated CNS infections may be considered once they resume baseline daily activities.
   2. Non-CNS opportunistic infections: Participants who recovered from or are completing treatment for non-CNS opportunistic infections (Ois) (e.g., Pneumocystis pneumonia, Candida esophagitis, or pulmonary TB) can be enrolled if they have returned to self-reported baseline activity and functional level.
2. Conditions other than HAND associated with cognitive impairment or dementia such as Alzheimer's, Parkinson's disease, head injury with loss of consciousness >30 minutes, untreated sleep apnea with day-time sleepiness, or seizure disorders. Participants with a history of seizure disorder with no seizure activity that are on a stable, non-sedating anti-seizure regimen for >6 months may be enrolled.
3. Concurrent severe, unstable psychiatric illness that, in the opinion of the investigators, may interfere with study participation and/or data interpretation. Participants on psychotropic anxiolytic, attention deficit-hyperactivity disorder (ADHD), and other psychiatric medications may be included if clinically stable for 6 months.
4. Concurrent substance abuse that, in the opinion of the investigators may interfere with study participation and/or data interpretation. Active substance abuse includes illegal drug use and/or excessive narcotic or alcohol use as determined by the investigator. Urine drug screen will be performed on all participants. Use of nicotine containing products will not be an exclusion criterion.
5. Contraindication to MRI scanning, including pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), implanted delivery pump, or shrapnel fragments. Participants requiring a low dose oral benzodiazepine for mild to moderate claustrophobia will be allowed to participate. Pregnancy testing will be performed in enrolled participants of childbearing potential 48 hours prior to any MRI.
6. Medications: narcotics, psychiatric, and anti-seizure medications will not be allowed except under certain conditions as noted above. Corticosteroids may be permitted for participants on stable short-term therapy without CNS disease (i.e. resolving Pneumocystis pneumonia). Participants must be willing not to take the following medications within 48 hours of neuropsychological testing: sedating antihistamines such as diphenhydramine, zolpidem and other drugs identified by the study team that are associated with altered alertness or impaired memory.
7. Prior or planned/anticipated exposure to radiation due to clinical care or participation in other research protocols, which would exceed the recommended acceptable annual limit of radiation exposure once accounting for the requirements of the current study.
8. Pregnant persons are excluded due to exposure to high magnetic fields There is also exposure to radiation from the lumbar puncture if done under fluoroscopy. Participants of childbearing potental must have a negative serum or urine pregnancy 48 hours prior to any radiation exposure.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any person meeting eligibility criteria and has no exclusionary criteria will be considered for the study.@@@
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2013-07-08 (Actual); Primary Completion 2037-02-22 (Estimated)

PRIMARY OUTCOMES:
To characterize in detail the natural course of HAND in subjects with prolonged plasma HIV virologic suppression (<50 copies/mL). | Annually
  The prevalence of neurocognitive impairment in this cohort will be high despite HIV plasma viremia below the limit of detection (BLD) in the blood as chronic activation may be mediating neuronal damage and result in cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antinori A, Arendt G, Becker JT, Brew BJ, Byrd DA, Cherner M, Clifford DB, Cinque P, Epstein LG, Goodkin K, Gisslen M, Grant I, Heaton RK, Joseph J, Marder K, Marra CM, McArthur JC, Nunn M, Price RW, Pulliam L, Robertson KR, Sacktor N, Valcour V, Wojna VE. Updated research nosology for HIV-associated neurocognitive disorders. Neurology. 2007 Oct 30;69(18):1789-99. doi: 10.1212/01.WNL.0000287431.88658.8b. Epub 2007 Oct 3. PMID 17914061
- [Background] McArthur JC. HIV dementia: an evolving disease. J Neuroimmunol. 2004 Dec;157(1-2):3-10. doi: 10.1016/j.jneuroim.2004.08.042. PMID 15579274
- [Background] Sacktor N, McDermott MP, Marder K, Schifitto G, Selnes OA, McArthur JC, Stern Y, Albert S, Palumbo D, Kieburtz K, De Marcaida JA, Cohen B, Epstein L. HIV-associated cognitive impairment before and after the advent of combination therapy. J Neurovirol. 2002 Apr;8(2):136-42. doi: 10.1080/13550280290049615. PMID 11935465
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-N-0149.html